CLINICAL TRIAL: NCT04161365
Title: Feasibility and Therapeutic Potential of Free Fat Grafts in the Treatment of Urethral Strictures
Acronym: UREGRAFT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hannes Kortekangas (Other Government)
Responsible Party: Sponsor-Investigator, Hannes Kortekangas, Gastrointestinal surgeon / Consultant in Division of Gastrointestinal Surgery, Turku University Hospital
Organization: Turku University Hospital (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UREGRAFT
Record Dates: First submitted 2019-07-29; First posted 2019-11-13 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Urethral Stricture; Fat Graft
Keywords: Urethral Stricture; Fat Graft; Direct Visual Urethrotomy
MeSH Terms: conditions — Urethral Stricture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Urethral stricture patients (Experimental): Patients suffering from urethral stricture are treated with direct visual internal urethrotomy (DVIU). Free fat graft is gathered from the abdominal subcutaneous fat. Fat graft is prepared and injected to the stricture site.
  Interventions: Procedure: Direct visual urethrotomy; Procedure: Autologous fat grafting

INTERVENTIONS:
Procedure: Direct visual urethrotomy — Urethral stricture is treated with urethrotomy under visual control
Procedure: Autologous fat grafting — Autologous fat graft is gathered and injected to stricture

SUMMARY:
In this study the investigators investigate the feasibility and therapeutic potential of free autologous fat grafting combined to direct visual urethrotomy (DVIU) in the treatment of urethral strictures.

DETAILED DESCRIPTION:
In this study the investigators wish to proof the concept of free fat grafting into urethral stricture via urethroscope. The investigators will recruit twenty male patients suffering from (endoscopy proven) benign stricture of spongy urethra. All recruited patients have undergone at least one direct visual internal urethrotomy (DVIU) before recruitment. IPSS-score and uroflowmetry are recorded upon recruitment. The IPSS-score is repeated one day preoperatively. Urine sample is gathered for bacterial and cytological analysis. Prophylactic single dose levofloxacin antibiotic is orally administered before operation.

The operation is performed in the operation room by one urologist and one surgeon under general anesthesia. First abdominal liposuction (roughly 20 ml) and fat graft preparation is performed. The fat graft is processed into nano-fat using Tulip GEMS Single-Use NanoTransfer Set. Then urethroscopy is performed, urethral stricture is visually graded (location, length, lumen), photographed, DVIU performed and nano fat graft (0,1-0,5ml) injected to stricture site beneath the mucosal layer at three locations. Urinary Foley ch 18 catheter is inserted. Patients are discharged the next day. Urinary catheter is removed after 20 hours.

Patients are contacted by phone 1 week after the operation. Post-operative symptoms are recorded and the patients are requested to contact the researcher if needed. Patient records are screened for pre- and postoperative symptoms, medication, long term illnesses and possible postoperative contacts to the hospital.

Three months later uroflowmetry, urethroscopy and IPSS-questionnaire are repeated. Stricture site is photographed and visually graded. In case of symptomatic re-stricture, the DVIU and fat grafting is repeated once. After 12 months uroflowmetry and IPSS-questionnaire are repeated. In case of suspected re-stricture the urethroscopy is repeated. Follow-up time is 12 months from the last fat graft injection.

Trial starts in fall 2019. The clinical studies have been completed and the data analysis and writing of the manuscript will be finalized in 2022.

ELIGIBILITY:
Inclusion Criteria:

* Urethral stricture that has re-occurred at least once.

Exclusion Criteria:

* Malignant etiology of urethral stricture

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-05-28 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events at 3 months | 3 months
  Types, severity and probability of procedure related adverse events
Incidence of Treatment-Emergent Adverse Events at 12 months | 12 months
  Types, severity and probability of procedure related adverse events

SECONDARY OUTCOMES:
Change from Baseline Uroflowmetry at 3 months | 3 months
  Measurements in uroflowmetry: Voided urine per unit of time, voided volume, maximum flow rate, curve of the flow.
Change from Baseline Uroflowmetry at 12 months | 12 months
  Measurements in uroflowmetry: Voided urine per unit of time, voided volume, maximum flow rate, curve of the flow.
Change from Baseline IPSS at 3 months | 3 months
  International Prostate Symptom Score (IPSS) is a validated symptom questionnaire used to measure voiding symptoms. Subscales: Incomplete emptying, frequency, intermittency, urgency, weak stream, straining, nocturia. Each sub scale 0-5 points. Zero points equal no symptoms and 5 points equal worst possible symptoms. Total 0-35 points.
Change from Baseline IPSS at 12 months | 12 months
  International Prostate Symptom Score (IPSS) is a validated symptom questionnaire used to measure voiding symptoms. Subscales: Incomplete emptying, frequency, intermittency, urgency, weak stream, straining, nocturia. Each sub scale 0-5 points. Zero points equal no symptoms and 5 points equal worst possible symptoms. Total 0-35 points.
Change from Baseline Stricture Lumen diameter at 3 months | 3 months
  Stricture photographed and lumen diameter measurement. Unit: closed biopsy forceps diameter.
Change from Baseline Stricture Lumen diameter at 12 months | 12 months
  Stricture photographed and lumen diameter measurement. Unit: closed biopsy forceps diameter.

CONTACTS AND LOCATIONS:
Overall Officials: Pauliina Hartiala, Surgeon, Study Director — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland